CLINICAL TRIAL: NCT02883699
Title: Individually Tailored Training Prescriptions in Cancer Patients: The TOP Study
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Friederike Rosenberger (University Hospital Heidelberg), Principal Investigator (Unknown); Dietmar Hopp Stiftung (Other)
Responsible Party: Principal Investigator, Joachim Wiskemann, Principle Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TOP-S-347/2016
Record Dates: First submitted 2016-08-16; First posted 2016-08-30 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Breast cancer; Prostate cancer; Exercise prescription; High intensity interval training; Daily undulating periodization training; Aerobic training; Resistance training; Physical fitness; Exercise
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Endurance Training Group 1 (Active Comparator): Standard endurance training
  Interventions: Behavioral: Standard endurance training
- Endurance Training Group 2 (Experimental): Polarized endurance training
  Interventions: Behavioral: Polarized endurance training
- Resistance Training Group 1 (Active Comparator): Standard resistance training
  Interventions: Behavioral: Standard resistance training
- Resistance Training Group 2 (Experimental): Daily undulating periodization resistance training
  Interventions: Behavioral: Daily undulating periodization resistance training

INTERVENTIONS:
Behavioral: Standard endurance training — Continuous vigorous training 2 x per week on a cycle ergometer
  Arms: Endurance Training Group 1
Behavioral: Polarized endurance training — Continuous moderate training 1 x per week and aerobic high intensity interval training (HIIT) 1 x per week on the cycle ergometer
  Arms: Endurance Training Group 2
Behavioral: Standard resistance training — Machine based hypertrophy training 2 x per week
  Arms: Resistance Training Group 1
Behavioral: Daily undulating periodization resistance training — Machine based daily undulating periodization resistance training 1 x per week
  Arms: Resistance Training Group 2

SUMMARY:
The TOP Study is a two-stage study on individually tailored endurance and resistance training prescriptions for breast and prostate cancer patients after the end of primary therapy in order to optimize training effects.

DETAILED DESCRIPTION:
The TOP Study is a two-stage study on individually tailored endurance and resistance training prescriptions for breast and prostate cancer patients after the end of primary therapy in order to optimize training effects.

The TOP Study Part I aims at identifying the most appropriate way of individual intensity prescription. In a descriptive cross sectional study, 20 breast and 20 prostate cancer patients perform singe endurance and resistance training sessions prescribed by means of different methods of intensity prescription. The most appropriate method of intensity prescription is identified through considering predictability/homogeneity of physiological responses as well as perceived exertion and enjoyment.

The TOP Study Part II aims at investigating the most effective training method in terms of enhancing physical fitness for both endurance and strength training. The design is an exploratory four-arm 12-week randomized controlled training intervention trial in 60 breast and 60 prostate cancer patients. In two endurance arms, vigorous continuous training is compared to a polarized program consisting of moderate training and aerobic high intensity interval training (HIIT). Similarly, in two resistance training arms, standard machine based hypertrophy training is compared to training following a daily undulating periodization design.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with early stage breast cancer (M0) or prostate cancer (M0 or M1 with PSA evidence of stable disease)
* 6 to 52 weeks after the end of primary therapy
* ≥18 to 75 years of age
* no regular endurance or resistance training (≥ one session per week) since diagnosis or within the last 6 months
* sufficient German language skills
* willing/ able to train at the provided exercise facilities twice per week and to take part in the scheduled testing
* signed informed consent.

Exclusion Criteria:

* diagnosed with additional other cancer
* brain or bone metastases in M1 prostate cancer patients
* heart failure >NYHA III, unstable angina pectoris or severe arrhythmia
* uncontrolled hypertension
* reduced standing or walking ability
* any other comorbidities that preclude participation in exercise testing or training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake (VO2peak) (endurance training groups only) | 12 weeks
  Change in maximal oxygen uptake (VO2peak) assessed in a maximal incremental exercise test (CPET) on a cycle ergometer
Change in one repetition maximum (1RM) of the knee extensors (resistance training groups only) | 12 weeks
  Change in one repetition maximum (1RM) of the knee extensors in a machine based 1RM test
Change in maximal isokinetic peak torque (MIPT) of the knee extensors (resistance training groups only) | 12 weeks
  Change in maximal isokinetic peak torque (MIPT) of the knee extensors assessed in a stationary dynamometer test

SECONDARY OUTCOMES:
Change in peak power output (PPO) (endurance training groups only) | 12 weeks
  Change in peak power output (PPO) assessed in a maximal incremental exercise test (CPET) on a cycle ergometer
Change in blood lactate threshold (endurance training groups only) | 12 weeks
  Change in blood lactate threshold assessed in a maximal incremental exercise test (CPET) on a cycle ergometer
Change in ventilatory threshold (endurance training groups only) | 12 weeks
  Change in ventilatory threshold assessed in a maximal incremental exercise test (CPET) on a cycle ergometer
Change in maximum voluntary isometric contraction (MVIC) of the knee extensors (resistance training groups only) | 12 weeks
  Change in maximum voluntary isometric contraction (MVIC) of the knee extensors assessed in a stationary dynamometer test
Change in total work (TW) of the knee extensors | 12 weeks
  Change in total work (TW) of the knee extensors assessed in a stationary dynamometer test
Change in muscular fatigue index (FI%) of the knee extensors | 12 weeks
  Change in muscular fatigue index (FI%) of the knee extensors assessed in a stationary dynamometer test
Adherence to the training programs | 12 weeks
  Adherence to the training programs
Drop-out rate in the training groups | 12 weeks
  Drop-out rate in the training groups
Pain during and between training sessions | 12 weeks
  Pain during and between training sessions (Brief Pain Inventory, BPI)
Minor and major adverse events during training sessions | 12 weeks
  Minor and major adverse events during training sessions
Changes in fatigue | 12 weeks
  Changes in fatigue (Multidimensional Fatigue Inventory, MFI 20)
Changes in Quality of Life (QoL) | 12 weeks
  Changes in Quality of Life (QoL) (European Research and Treatment in Cancer Quality of Life Questionnaire, EORTC QLQ-C30)
Changes in depression | 12 weeks
  Changes in depression (Center for Epidemiologic Studies Depression Scale, CES-D)
Enjoyment of the training programs | 12 weeks
  Enjoyment of the training programs (according to Rogers)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, Dr., Principal Investigator — Heidelberg University Hospital, National Center for Tumor Diseases, Division of Medical Oncology, Working Group Exercise Oncology
Locations (1):
- Heidelberg University Clinic, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelzer F, Leisge K, Schluter K, Schneider J, Wiskemann J, Rosenberger F. Effects of exercise mode and intensity on patient-reported outcomes in cancer survivors: a four-arm intervention trial. Support Care Cancer. 2023 May 2;31(5):315. doi: 10.1007/s00520-023-07757-9. PMID 37129687